CLINICAL TRIAL: NCT01702909
Title: Phase II Trial of Moderate Dose Bolus Interleukin-2 in Metastatic Kidney Cancer
Brief Title: Interleukin-2 in Metastatic Kidney Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: PI Decision
Sponsor: Western Regional Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-08
Record Dates: First submitted 2012-10-04; First posted 2012-10-10 (Estimated); Results first posted 2017-09-27 (Actual); Last update posted 2018-02-08 (Actual); Status verified 2018-02

CONDITIONS: Renal Cell Cancer Metastatic; Kidney Cancer Metastatic
Keywords: Metastatic Renal Cell; Metastatic Kidney Cancer
MeSH Terms: conditions — Kidney Neoplasms | interventions — Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Interleukin-2 (Experimental): Interleukin-2
  Interventions: Drug: Interleukin-2

INTERVENTIONS:
Drug: Interleukin-2 — Interleukin-2
  Other Names: IL2

SUMMARY:
The purpose of this study is to determine whether Interleukin-2 at the dose and schedule used in this study will help increase tumor shrinkage.

DETAILED DESCRIPTION:
In this phase II study, the IL-2 schedule (daily IL-2 for 5 days (per week) every 3 weeks) will be tested in a cohort of kidney cancer patients to attempt to determine the response rate, median duration of response, and median survival. The dose intensity of this schedule would allow a patient treated on this regimen to achieve the target threshold (> 1440 million IU/m2/year).

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have a histologic diagnosis of metastatic kidney cancer. Patients may have received prior systemic therapy or may be previously untreated
2. Patients must have bi-dimensional measurable disease on physical exam or radiologic studies.
3. ECOG performance status of 0 or 1 and estimated survival of at least 3 months.
4. White blood count of > 3500/mm3, platelet count > 100,000/mm3, hemoglobin > 9.0 gm/dl; bilirubin, ALT, AST < 3 x upper limit of normal; serum creatinine < 2.0 mg/dl.
5. Patients must undergo a low-level cardiac stress test as a screen for possible atherosclerotic heart disease. Patients with a positive stress test would be excluded from this trial.
6. Patients with elevated temperatures > 100.5 F must have sources of occult infection excluded.
7. Patients must be felt to have recovered from effects of prior therapy, such as > 2 weeks after prior chemotherapy.
8. Patient consent must be obtained prior to entrance onto study.
9. Women of childbearing potential must have a negative pregnancy test and must take adequate precautions to prevent pregnancy during treatment

Exclusion Criteria:

1. Medical illness requiring corticosteroids or other immunosuppressive agents (such as cyclosporin or methotrexate.
2. Autoimmune disease such as inflammatory arthritis which could be exacerbated by immune-based therapy.
3. Prior history of psychiatric disorder which could be exacerbated by interleukin-2.
4. Lactation or pregnancy.
5. Evidence of significant cardiovascular disease including history of recent (< 6 months prior) myocardial infarction, congestive heart failure, primary cardiac arrhythmias (not due to electrolyte disorder or drug toxicity, for example) beyond occasional PVC's, angina, positive low-level stress test, or cerebrovascular accident.
6. Current brain metastasis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2012-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Quan, MD, Principal Investigator — Western Regional Medical Center
Locations (1):
- Western Regional Medical Center, Inc, Goodyear, Arizona, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Interleukin-2: Interleukin 2 (IL-2) is naturally produced by the body to help fight infection and prevent autoimmune diseases. In cancer treatment, IL-2 is designed to target adaptive immune cells, such as T-cells and B-cells, to respond to tumors. IL-2 may help the body produce antigen-fighting T-cells and stimulate B-cells to produce more antibodies.
Period: Overall Study
Arm/Group | Interleukin-2
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Number of Participants: Treated with Interleukin-2
Arm/Group | Number of Participants
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Age, Continuous [Median (Full Range); unit: years] | 58 [54 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Response Using RECIST Criteria
Description: Radiographic studies to evaluate for response were done after every 2 cycles (6 weeks) until disease progression or death from any cause up to 2 years. Standard RECIST response criteria were utilized. Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by CT scan: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response Rate (ORR) = 100%(CR + PR/total number of patients receiving Interleukin-2).
Time Frame: Measured until Disease Progression or death from any cause up to 2 year
Population: No data was collected
Groups:
- Response Rate: Percentage of Patients Responding to Interleukin-2
Arm/Group | Response Rate
Number analyzed (Participants) | 0

2. Secondary Outcome: Median Duration of Response
Description: Duration of response is calculated as the time (months) from the date at which response is first observed (per standard Response Evaluation Criteria In Solid Tumors [RECIST] to the date of first observed disease progression or date of death from any cause, whichever came first, assessed up to 2 years. The actual date of tumor assessments was used for this calculation. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of one or more new lesions.
Time Frame: Measured from first response until Disease Progression or death from any cause up to 2 years
Population: There are no data recordings for this study. The study was terminated and the investigator is no longer related to the site. There is no additional information to provide.
Arm/Group | Response Rate
Number analyzed (Participants) | 0

3. Secondary Outcome: Median Survival
Description: from time of study entry until death
Time Frame: measured from date of first dose until date of death
Population: as for outcome 2
Arm/Group | Response Rate
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Through study completion, approximately 2 years
Groups:
- Adverse Events: Patients receiving Interleukin-2
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 7/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 7/7
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Adverse Events (N=7)
Nausea/emesis (Gastrointestinal disorders) | 7
Decreased appetite (Metabolism and nutrition disorders) | 6
Rigors (General disorders) | 6
Catarrhal/sinus symptoms (General disorders) | 5
Constipation (Gastrointestinal disorders) | 4
Arthalgia/myalgia (Musculoskeletal and connective tissue disorders) | 4
Fever (General disorders) | 4
Peripheral swelling (General disorders) | 4
Skin rash (Skin and subcutaneous tissue disorders) | 3
Headache (Nervous system disorders) | 3
Elevated creatinine (Investigations) | 2
Fatigue (General disorders) | 2
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes